CLINICAL TRIAL: NCT02832375
Title: A Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Brief Title: Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205697
Record Dates: First submitted 2016-03-28; First posted 2016-07-14 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: stannous fluoride (Experimental): Participants will be instructed to dose a dry toothbrush containing 0.454% w/w of stannous fluoride (1000 parts per million [ppm] fluoride) with a full strip (1 inch) of toothpaste. Participants will then brush each of the two selected sensitive test teeth first followed by the whole mouth thoroughly for at least 1 minute.
  Interventions: Drug: stannous fluoride
- Standard: sodium monofluorophosphate (Active Comparator): Participants will be instructed to dose a dry toothbrush containing 0.76% w/w sodium monofluorophosphate (1000ppm fluoride) with a full strip (1 inch) of toothpaste. Participants will then brush each of the two selected sensitive test teeth first followed by the whole mouth thoroughly for at least 1 minute.
  Interventions: Drug: sodium monofluorophosphate

INTERVENTIONS:
Drug: stannous fluoride — 0.454% w/w stannous fluoride containing 1100ppm of fluoride
  Arms: Experimental: stannous fluoride
Drug: sodium monofluorophosphate — 0.76% w/w sodium monofluorophosphate containing 1000ppm fluoride
  Arms: Standard: sodium monofluorophosphate

SUMMARY:
This single center, comparative design study will be used to investigate the efficacy of an experimental stannous fluoride containing dentifrice in relieving dentinal hypersensitivity (DH) after short term use compared with a standard fluoride dentifrice.

DETAILED DESCRIPTION:
This will be a single center, three day, randomized, examiner blind, two treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected test teeth), controlled study, in participants with at least two sensitive teeth that meet all the criteria at the screening and baseline (pre-treatment) visits. DH will be assessed at baseline (pre-treatment), post-treatment and after 3 days twice daily brushing.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged 18-65 years inclusive
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant, relevant abnormalities of medical history or oral examination and Absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements
* Self-reported history of DH lasting more than six months but not more than 10 years at screening
* Minimum of 20 natural teeth at screening
* Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants that meet all of the following criteria: Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR) Tooth with MGI score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of less than or equal to (≤)1 and Tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y[Yes]/N[No] response) screening
* Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars),that meet all of the following criteria at Baseline: Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff sensitivity score ≥ 2)

Exclusion Criteria:

* Women who are known to be pregnant. Females of child bearing potential who have a positive urine pregnancy test or who are breast feeding
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Previous participation in this study or participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit
* Recent history (within the last year) of alcohol or other substance abuse
* An employee of the sponsor or the study site or members of their immediate family
* Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes or Any condition which, in the opinion of the investigator, causes xerostomia
* Dental prophylaxis within 4 weeks of Screening, tongue or lip piercing or presence of dental implants, gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening and teeth bleaching within 8 weeks of Screening
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine
* Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the Investigator
* Use of an oral care product indicated for the relief of dentine hypersensitivity within 8 weeks of screening
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, anti-depressants, mood-altering and anti-inflammatory drugs.
* Currently taking antibiotics or has taken antibiotics within 2 weeks of Baseline, Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-03-01; Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Creeth J, Gallob J, Sufi F, Qaqish J, Gomez-Pereira P, Budhawant C, Goyal C. Randomised clinical studies investigating immediate and short-term efficacy of an occluding toothpaste in providing dentine hypersensitivity relief. BMC Oral Health. 2019 Jun 4;19(1):98. doi: 10.1186/s12903-019-0781-x. PMID 31164116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one center in United States.
Pre-assignment Details: A total of 266 participants were screened, out of which 242 participants were randomized. 24 participants were not randomized because 14 participants did not met the study criteria, 1 participant was lost to follow up and 9 participants withdrew consent from the study.
Groups:
- Experimental: Stannous Fluoride(SnF): Participants were instructed to dose a dry toothbrush containing 0.454% weight by weight (w/w) of SnF (1100 parts per million [ppm] fluoride) with a full strip (1 inch) of toothpaste. Participants then brushed each of the two selected sensitive test teeth first followed by the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
- Control: Sodium Monofluorophosphate(SMFP): Participants were instructed to dose a dry toothbrush containing 0.76% w/w SMFP (1000ppm fluoride) with a full strip (1 inch) of toothpaste. Participants then brushed their whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
Period: Overall Study
Arm/Group | Experimental: Stannous Fluoride(SnF) | Control: Sodium Monofluorophosphate(SMFP)
Started | 121 | 121
Completed | 119 | 121
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal of Consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Stannous Fluoride(SnF): Participants were instructed to dose a dry toothbrush containing 0.454% w/w of SnF (1100ppm fluoride) with a full strip (1 inch) of toothpaste. Participants then brushed each of the two selected sensitive test teeth first followed by the whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
- Total: Total of all reporting groups
Arm/Group | Experimental: Stannous Fluoride(SnF) | Control: Sodium Monofluorophosphate(SMFP) | Total
Number analyzed (Participants) | 121 | 121 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (11.32) | 37.4 (11.01) | 37.7 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 78 | 154
  Male | 45 | 43 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 19 | 46
  Not Hispanic or Latino | 94 | 102 | 196
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 25 | 27 | 52
  White | 74 | 72 | 146
  More than one race | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Shiff Sensitivity Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Assessed by examiner as participant's response to an evaporative (air) stimulus after stimulation of each individual tooth, scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus & requests discontinuation or moves from stimulus; 3=Participant responds to stimulus, considers stimulus to be painful, & requests discontinuation of stimulus. A reduction in Schiff Sensitivity score indicates improvement in sensitivity. Population: This baseline measurement was performed on intent-to-treat (ITT) population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy.
  score on a scale | 2.53 (0.389) | 2.55 (0.397) | 2.54 (0.392)
Tactile Threshold at Baseline [Mean (Standard Deviation); unit: gram (g)] — Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 g to an upper threshold of 80g in increments of 10 g. Tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. Tactile threshold for each tooth was determined by asking participant whether sensation caused discomfort. The pressure setting at which participant gave two consecutive 'yes' responses was recorded as tactile threshold. Higher tactile threshold, less sensitive tooth. Population: This baseline measurement was performed on ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy.
  gram (g) | 10.00 (0.000) | 10.00 (0.000) | 10.00 (0.000)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 3
Description: Schiff sensitivity score was assessed by examiner as participant's response to an evaporative (air) stimulus after the stimulation of each individual tooth. Response of participant was scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3= Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score indicates improvement in sensitivity.
Time Frame: Baseline, Day 3
Population: Analysis for this outcome was conducted on ITT population, defined as all participants who were randomized, received study treatment at least once & provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed is number of participants from ITT population evaluated on Day 3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Stannous Fluoride(SnF) | Control: Sodium Monofluorophosphate(SMFP)
Number analyzed (Participants) | 119 | 121
score on a scale | -0.82 (0.644) | -0.39 (0.426)
Statistical Analysis 1: Comparison: Experimental: Stannous Fluoride(SnF) vs Control: Sodium Monofluorophosphate(SMFP); H0= no difference between experimental dentifrice and control dentifrice H1= a difference between experimental dentifrice and control dentifrice; Test type: Superiority or Other; p < 0.0001, ANCOVA; From ANCOVA model with change from baseline in Schiff Sensitivity Score as response and treatment and baseline Schiff sensitivity score as covariates; Least Square (LS) mean difference = -0.45, 95% CI 2-sided [-0.577 to -0.319] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favours first named dentifrice

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score After Single Use
Description: as for outcome 1
Time Frame: Baseline, after single use (after 5 minutes)
Population: Analysis for this outcome was conducted on ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment of efficacy. Number of participants analyzed is the ITT Population evaluated post treatment single usage for each treatment arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standard: Sodium Monofluorophosphate(SMFP): Participants were instructed to dose a dry toothbrush containing 0.76% w/w SMFP (1000ppm fluoride) with a full strip (1 inch) of toothpaste. Participants then brushed their whole mouth thoroughly for at least 1 minute. Participants were permitted to rinse with tap water after brushing.
Arm/Group | Experimental: Stannous Fluoride(SnF) | Standard: Sodium Monofluorophosphate(SMFP)
Number analyzed (Participants) | 121 | 121
score on a scale | -0.46 (0.507) | -0.45 (0.465)

3. Secondary Outcome: Change From Baseline in Tactile Threshold Immediately After Single Use and on Day 3
Description: Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 g to an upper threshold of 80g in increments of 10 g. The tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gave two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth.
Time Frame: Baseline, after single use (after 5 minutes) and on Day 3
Population: Analysis for this outcome was conducted on ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment of efficacy. n=number of participants evaluated at specific time points for each treatment arms respectively.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Experimental: Stannous Fluoride(SnF) | Standard: Sodium Monofluorophosphate(SMFP)
Number analyzed (Participants) | 121 | 121
g
  Change from baseline post treatment | 4.01 (7.545) | 3.60 (7.252)
  Change from baseline on Day 3: number analyzed (Participants) | 119 | 121
  Change from baseline on Day 3 | 15.25 (17.766) | 3.88 (6.785)

ADVERSE EVENTS:
Arm/Group | Experimental: Stannous Fluoride(SnF) | Standard: Sodium Monofluorophosphate(SMFP)
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/121
Other Adverse Events (participants affected / at risk) | 1/121 | 2/121
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Stannous Fluoride(SnF) (N=121) | Standard: Sodium Monofluorophosphate(SMFP) (N=121)
Oral Mucosal Exfoliation (Gastrointestinal disorders) | 1 | 0
Leukoplakia Oral (Gastrointestinal disorders) | 0 | 1
Lip Ulceration (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.